CLINICAL TRIAL: NCT03845361
Title: Does Radial Artery Cannulation Affect the Perfusion of the Dominant Hand in Patients Undergoing Open Cardiac Surgery? Data Derived From the Peripheral Perfusion Index.
Brief Title: Radial Artery Cannulation and Perfusion Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Radial perfusion index
Record Dates: First submitted 2018-12-25; First posted 2019-02-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Perfusion
Keywords: Perfusion index; Cardiac Surgery; Radial artery cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C. hand (Experimental): Radial artery cannulation
  Interventions: Procedure: Radial artery cannulation
- N.C. hand (No Intervention): No cannulation of the radial artery

INTERVENTIONS:
Procedure: Radial artery cannulation — Radial artery cannulation
  Arms: C. hand

SUMMARY:
This study aims to investigate if radial artery cannulation of the dominant hand affects its peripheral perfusion during cardiac surgery using cardiopulmonary bypass.

DETAILED DESCRIPTION:
Invasive blood pressure monitoring is mandatory in cardiac surgeries. Radial artery cannulation is the most common technique used for monitoring of invasive blood pressure and for arterial blood gas analysis.

Perfusion index derived from pulse oximetry is a new method for monitoring of peripheral perfusion.

this study aims to investigate if radial artery cannulation affects the intra-operative peripheral perfusion in the dominant cannulated hand

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* Peripheral vascular diseases
* previous upper limb surgeries
* planned radial artery harvesting

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
The perfusion index | Intraoperative
The peripheral temperature | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided